CLINICAL TRIAL: NCT00621361
Title: A Phase I, Multi-Centre, Open-Label, Dose Selection Study to Assess the Safety and Tolerability of Cediranib (RECENTIN™, AZD2171) in Combination With Etoposide and Cisplatin (EP) as First Line Therapy for Lung Cancer Patients With Extensive Stage or Metastatic Disease for Whom EP Would be a Standard Therapy
Brief Title: Phase I Safety and Tolerability Study of Cediranib (RECENTIN™, AZD2171) in Combination With Chemo in First Line Lung Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00054
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; AZD2171; cediranib; RECENTIN; etoposide; cisplatin
MeSH Terms: conditions — Lung Neoplasms | interventions — cediranib; Etoposide; etoposide phosphate; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD2171
- 2 (Active Comparator): Etoposide + Cisplatin
  Interventions: Drug: Etoposide; Drug: Cisplatin

INTERVENTIONS:
Drug: AZD2171 — Oral
  Other Names: Recentin™
  Arms: 1
Drug: Etoposide — Intravenous
  Other Names: Etopophos®
  Arms: 2
Drug: Cisplatin — Intravenous
  Other Names: Platinol
  Arms: 2

SUMMARY:
This study is to assess the safety and tolerability of Cediranib (RECENTIN™, AZD2171)in combination with etoposide and cisplatin (EP) as first line treatment for lung cancer patients with extensive stage or metastatic disease for whom EP would be a standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis and stage (histological or cytological confirmed extensive stage lung cancer, which EP would be considered a standard therapy, required at the time of diagnosis.)
* No prior chemotherapy or immunotherapy for advanced stage lung cancer (prior radiotherapy will be permitted if it is outside of the measurable field and greater than or equal to 2 weeks prior to entry to the study.)
* WHO performance status 0-2

Exclusion Criteria:

* Untreated unstable brain or meningeal metastases
* Patient with inappropriate laboratory tests values
* Inadequate bone marrow reserve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of Cediranib (RECENTIN™, AZD2171) in combination with etoposide and cisplatin (EP). | From date of consent through to data cut-off, 7th August 2009.

SECONDARY OUTCOMES:
Preliminary efficacy assessment of Cediranib in combination with etoposide & cisplatin using available tumor assessment data to assess response rate,duration of response,change in tumor size(only those with measurable disease)& progression free survival | From date of randomisation through to data cut-off, 7th August 2009.

CONTACTS AND LOCATIONS:
Overall Officials: John Heymach, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Research Site, Sacramento, California
  - Research Site, Denver, Colorado
  - Research Site, Kansas City, Kansas
  - Research Site, Houston, Texas